CLINICAL TRIAL: NCT01571427
Title: Conversational Engagement as a Means to Delay Alzheimer's Disease Onset
Brief Title: Conversations as a Means to Delay the Onset of Alzheimer's Disease
Acronym: conversation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Hiroko H. Dodge, Professor of Neurology, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: socialengagementR01; R01AG033581 (NIH)
Record Dates: First submitted 2012-03-29; First posted 2012-04-05 (Estimated); Results first posted 2019-04-24 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Mild Cognitive Impairment; Cognitive Change
Keywords: Behavioral intervention; Social engagement; Conversational engagement; Social network; Cognitive Reserve; Alzheimer's disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Experimental and control groups. The experimental group will have 30 minutes daily (5 times per week) video chat with standardized conversational staff for 6 weeks, while the control group will have phone check-in once per week for 10 minutes for increasing retention. Both groups will complete weekly web-based heath form using PC and internet.
Who Masked: Outcomes Assessor
Masking Description: Investigators and assessors are blind to the group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): No daily conversational sessions with interviewers using webcam/internet. Weekly web-based heath form must be submitted using internet/PC. If not, subjects receive prompts from study personnel.
  Interventions: Behavioral: Control group
- Active social engagement group (Active Comparator): Engage in 30 minutes video chat daily (5 times per week, except weekend) with interviewers for 6 weeks. Weekly web-based heath form must be submitted using internet/PC. If not, subjects receive prompts from study personnel.
  Interventions: Behavioral: Active social engagement group

INTERVENTIONS:
Behavioral: Active social engagement group — Engage in 30 minutes conversation daily using internet/webcam, 5 days per week for 6 weeks, tracking of daily conversational amount outside of the trial by using a digital recording device, lasting effects will be assessed at the 3rd and 6th month after completion of the intervention
  Arms: Active social engagement group
Behavioral: Control group — No active intervention, weekly phone calls by interviewer to complete health/social engagement monitoring survey, tracking of daily conversational amount by using a digital recording device. Participants will be reassessed at the 3rd and 6th month after completion of the intervention.
  Arms: Control group

SUMMARY:
Past epidemiological studies have demonstrated that larger social networks, or more frequent social interactions, could have potential protective effects on the incidence of Alzheimer's Disease (AD). However, in those studies, indicators of social interactions were often broad, and included distinct elements that affected cognition and overall health. This project will examine whether conversation-based cognitive stimulation has positive effects on domain-specific cognitive functions among the elderly. Face-to-face communication will be conducted through the use of personal computers, webcams, and user-friendly simple interactive Internet programs to allow participants to have social engagement while staying at their home and also for the cost effective execution of the study.

DETAILED DESCRIPTION:
Participants are randomized into the control group (weekly 10 minutes phone check-in only) or experimental group (30 minutes daily video chat with standardized/trained conversational staff). User-friendly equipment and internet are provided.

ELIGIBILITY:
Inclusion Criteria:

* Non-demented participants
* Willing to participate in daily conversation using internet/webcam with interviewers for 6 weeks
* Willing to monitor daily conversational amount using a digital recording device
* Willing informant who has frequent contact with the participant

Exclusion Criteria:

* have major illness or disabilities which interfere with interacting using the audio/video technology
* diagnosed as dementia
* MMSE < 24 at screening
* Geriatric Depression Scale (15 items) >4 at screening

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 83 (Actual)
Dates: Start 2012-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided
completely de-identified data are available upon requests

REFERENCES:
- [Background] Dodge HH, Katsumata Y, Zhu J, Mattek N, Bowman M, Gregor M, Wild K, Kaye JA. Characteristics associated with willingness to participate in a randomized controlled behavioral clinical trial using home-based personal computers and a webcam. Trials. 2014 Dec 23;15:508. doi: 10.1186/1745-6215-15-508. PMID 25539637
- [Background] Asgari M, Kaye J, Dodge H. Predicting mild cognitive impairment from spontaneous spoken utterances. Alzheimers Dement (N Y). 2017 Feb 27;3(2):219-228. doi: 10.1016/j.trci.2017.01.006. eCollection 2017 Jun. PMID 29067328
- [Background] Dodge HH, Mattek N, Gregor M, Bowman M, Seelye A, Ybarra O, Asgari M, Kaye JA. Social Markers of Mild Cognitive Impairment: Proportion of Word Counts in Free Conversational Speech. Curr Alzheimer Res. 2015;12(6):513-9. doi: 10.2174/1567205012666150530201917. PMID 26027814
- [Result] Dodge HH, Zhu J, Mattek N, Bowman M, Ybarra O, Wild K, Loewenstein DA, Kaye JA. Web-enabled Conversational Interactions as a Means to Improve Cognitive Functions: Results of a 6-Week Randomized Controlled Trial. Alzheimers Dement (N Y). 2015 May;1(1):1-12. doi: 10.1016/j.trci.2015.01.001. PMID 26203461
- [Result] Cerino ES, Hooker K, Goodrich E, Dodge HH. Personality Moderates Intervention Effects on Cognitive Function: A 6-Week Conversation-Based Intervention. Gerontologist. 2020 Jul 15;60(5):958-967. doi: 10.1093/geront/gnz063. PMID 31112605
- See also: Web-enabled conversational interactions as a means to improve cognitive functions: Results of a 6-week randomized controlled trial — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4507295/
- See also: Characteristics associated with willingness to participate in a randomized controlled behavioral clinical trial using home-based personal computers and a webcam — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4307639/
- See also: Predicting mild cognitive impairment from spontaneous spoken utterances — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5651423/
- See also: Social markers of mild cognitive impairment: Proportion of word counts in free conversational speech — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4526336/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From November 2011 to August 2012, we distributed 2000 surveys targeting those living in retirement communities and senior centers located in the Portland, metropolitan area, within an approximately 1-hour commute from Oregon Health & Science University (Portland, OR).
Groups:
- Active Social Engagement Group: Active Social Engagement: Engage in 30 minutes conversation daily with interviewers using internet/webcam for 6 weeks
  Active social engagement group: Engage in 30 minutes conversation daily using internet/webcam, 5 days per week for 6 weeks, tracking of daily conversational amount outside of the trial by using a digital recording device, lasting effects will be assessed at the 3rd and 6th month after completion of the intervention
- Control Group: No daily conversational sessions with interviewers using webcam/internet. Weekly web-based heath form must be submitted using internet/PC. If not, subjects receive prompts from study personnel.
  Control group: No active intervention, weekly phone calls by interviewer to complete health/social engagement monitoring survey, tracking of daily conversational amount by using a digital recording device
Period: Overall Study
Arm/Group | Active Social Engagement Group | Control Group
Started | 41 | 42
Completed | 41 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Active Soocial Engagement Group: Active Social Engagement: Engage in 30 minutes conversation daily with interviewers using internet/webcam for 6 weeks
  Active social engagement group: Engage in 30 minutes conversation daily using internet/webcam, 5 days per week for 6 weeks, tracking of daily conversational amount outside of the trial by using a digital recording device, lasting effects will be assessed at the 3rd and 6th month after completion of the intervention
- Total: Total of all reporting groups
Arm/Group | Active Soocial Engagement Group | Control Group | Total
Number analyzed (Participants) | 41 | 42 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.9 (7.2) | 80.2 (6.6) | 80.5 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 31 | 63
  Male | 9 | 11 | 20
Region of Enrollment [Number; unit: participants]
  United States | 41 | 42 | 83
Education: High school completed or greater [Count of Participants; unit: Participants] | 40 | 40 | 80
Cognitive Status: Clinical Dementia Rating (CDR) Scale score of 0.5 (%) [Count of Participants; unit: Participants] — Range (0, 0.5) CDR=0 is operationally defined as having normal cognition. CDR=0.5 is operationally defined as having Mild Cognitive Impairment (MCI)
  Participants | 17 | 17 | 34
Global cognitive Status: Mini-Mental State Examination score [Mean (Standard Deviation); unit: units on a scale] — Global cognitive function score (possible score ranges from 0 to 30). In this study, score ranges from 24 to 30 (those with MMSE<24 were excluded according to the study exclusion criteria). Higher score indicates better cognitive function.
  units on a scale | 28.2 (1.7) | 28.3 (1.8) | 28.3 (1.8)
Marital Status: Married (%) [Count of Participants; unit: Participants] | 18 | 20 | 38
Levels of Education: The Wide Range Achievement Test--Revised (WRAT-R) [Mean (Standard Deviation); unit: units on a scale] — The Wide Range Achievement Test--Revised (WRAT-R). Score ranges from 0 to 89. Higher score indicate better reading ability.
  units on a scale | 72.0 (12.9) | 72.0 (11.5) | 72.0 (12.1)
Experience using personal computer (PC) [Count of Participants; unit: Participants] | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Changes in Global Cognitive Function Using Mini Mental State Examination Score (Post-study Test Score - Baseline Test Score)
Description: Mini Mental State Examination assess global cognitive function. Possible score ranges from 0 to 30. In this study, score ranges from 24 to 30 (those with MMSE <24 at baseline were excluded according to the study exclusion criteria). Changes in test results among the experimental group are compared with changes among the control group using linear regression models. (no drop out reported and therefore no need to use mixed effects models or MMRM) Higher values (post-pre) indicate that decline was less or test score improved more.
Time Frame: 6 weeks (primary endpoint) from baseline
Population: Sampling frame consists of retirement communities and Layton Aging Alzheimer's Disease research center volunteer lists. The survey asking whether they would like to participate in the study was distributed among 2000 subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Social Engagement Group | Control Group
Number analyzed (Participants) | 41 | 42
score on a scale | -0.51 (1.51) | -0.07 (1.65)
Statistical Analysis 1: Comparison: Active Social Engagement Group vs Control Group; Test type: Equivalence — It was calculated that 82 participants randomized in a 1:1 fashion between the 2 arms would have at least 80% to detect a Cohen's D of 0.45 in the difference in changes from baseline to week 6 at alpha=0.05 (two tailed). All randomized participants (n=83) were included in the analysis; p = 0.25, Regression, Linear; Mean Difference (Final Values) = -0.41, Standard Error of Mean 0.35 — Estimates reported here is coefficient for the experimental group (with the control group as a reference), using a linear regression model controlling for Geriatric Depression Scale - 15 items version (GDS-15)
Statistical Analysis 2: Comparison: Active Social Engagement Group vs Control Group; Analysis 2: AMONG CDR=0 group (N=49); Test type: Equivalence — Power calculation was based on the entire sample (CDR=0 and CDR=0.5 combined). Analyses within each CDR group are exploratory; p = 0.25, Regression, Linear; Median Difference (Final Values) = -0.49, Standard Error of Mean 0.42 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Active Social Engagement Group vs Control Group; Analyses 3: AMONG CDR=0.5 (Mild Cognitive Impairment) group, N=34; Test type: Equivalence — Power calculation was based on the entire sample which combined CDR=0 and CDR=0.5 groups. Analyses within each CDR group are exploratory; p = 0.85, Regression, Linear; Median Difference (Final Values) = -0.11, Standard Error of Mean 0.62 — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Changes in Category Fluency (Animals) Test Scores (Post-study Test Score - Baseline Test Score)
Description: Verbal fluency Animals test is a neuropsychological test. In the test, participants have to produce as many words as possible from a category of animals within 60 seconds. Total score ranges from 0 to 70. Changes in test results among the experimental group are compared with changes among the control group using linear regression models. (no drop out reported and therefore no need to use mixed effects models or MMRM). Higher values mean decline is less or score improve at post-study assessment.
Time Frame: 6 weeks (primary endpoint) from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of words
Arm/Group | Active Social Engagement Group | Control Group
Number analyzed (Participants) | 41 | 42
Number of words | 1.75 (4.21) | -0.38 (4.08)
Statistical Analysis 1: Comparison: Active Social Engagement Group vs Control Group; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.02, Regression, Linear; Mean Difference (Final Values) = 2.20, Standard Error of Mean 0.92 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Active Social Engagement Group vs Control Group; Analysis 2: AMONG CDR=0 group (N=49); Test type: Equivalence — Power calculation was based on the entire sample which combined CDR=0 and CDR=0.5 groups. Analyses by each CDR group are exploratory; p = 0.003, Regression, Linear — Statistically significant based on the Bonferroni multiple comparison adjusted P value of P<0.004; Mean Difference (Final Values) = 4.00, Standard Error of Mean 1.28 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Active Social Engagement Group vs Control Group; Analyses 3: CDR=0.5 (Mild Cognitive Impairment) group, N=34; Test type: Equivalence — [test comment as in outcome 2, analysis 2]; p = 0.65, Regression, Linear; Mean Difference (Final Values) = 0.52, Standard Error of Mean 1.14 — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Changes in Verbal Fluency Letter Test Scores (Post-study Test Score - Baseline Test Score)
Description: Verbal fluency letter test is a neuropsychological test. In the test, participants have to produce as many words as possible which start with a letter F, A and S (3 separate test for each letter) within 60 seconds. Each test score ranges from 0 to 40. Total of 3 tests scores (F, A and S) ranges from 0 to 120. Changes in test results among the experimental group are compared with changes among the control group using linear regression models. (no drop out reported and therefore no need to use mixed effects models or MMRM) Higher values mean decline is less or test scores improved at post-study assessment.
Time Frame: 6 weeks (primary endpoint) from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of words
Arm/Group | Active Social Engagement Group | Control Group
Number analyzed (Participants) | 41 | 42
Number of words | 1.14 (6.45) | 1.26 (5.59)
Statistical Analysis 1: Comparison: Active Social Engagement Group vs Control Group; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.98, Regression, Linear; Mean Difference (Final Values) = 0.03, Standard Error of Mean 1.33 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Active Social Engagement Group vs Control Group; Analysis 2: Among CDR 0 (n=49); Test type: Equivalence — [test comment as in outcome 2, analysis 2]; p = 0.96, Regression, Linear; Mean Difference (Final Values) = -0.09, Standard Error of Mean 1.63 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Active Social Engagement Group vs Control Group; Analysis 3: Among CDR 0.5 (n=34); Test type: Equivalence — [test comment as in outcome 2, analysis 2]; p = 0.83, Regression, Linear; Mean Difference (Final Values) = 0.51, Standard Error of Mean 2.38 — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Changes in the Consortium to Establish a Registry for Alzheimer's Disease Word List Immediate Recall (Post-study Test Score - Baseline Test Score)
Description: Consortium to Establish a Registry for Alzheimer's Disease Word List Immediate Recall (CERAD Word List Immediate Recall) total score counts number of words correctly recalled over 3 trials (with each trial having 10 words), and ranges from 0 to 30. Pre-post changes in test results among the experimental group were compared with pre-post changes among the control group using linear regression models. (no drop out reported and therefore no need to use mixed effects models or MMRM)
Time Frame: 6 weeks (primary endpoint) from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of words
Arm/Group | Active Social Engagement Group | Control Group
Number analyzed (Participants) | 41 | 42
Number of words | 0.30 (2.69) | 0.53 (3.03)
Statistical Analysis 1: Comparison: Active Social Engagement Group vs Control Group; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.68, Regression, Linear; Mean Difference (Final Values) = -0.27, Standard Error of Mean 0.64 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Active Social Engagement Group vs Control Group; Analysis 2: CDR 0 (n=49); Test type: Equivalence — [test comment as in outcome 2, analysis 2]; p = 0.69, Regression, Linear; Mean Difference (Final Values) = -0.34, Standard Error of Mean 0.84 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Active Social Engagement Group vs Control Group; Analysis 3: CDR 0.5 (n=34); Test type: Equivalence — [test comment as in outcome 2, analysis 2]; p = 0.86, Regression, Linear; Mean Difference (Final Values) = -0.18, Standard Error of Mean 1.02 — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: Changes in the Consortium to Establish a Registry for Alzheimer's Disease Word List Delayed Recall (Post-study Test Score - Baseline Test Score)
Description: Consortium to Establish a Registry for Alzheimer's Disease Word List Delayed Recall (CERAD Word List Delayed Recall) total score counts number of words correctly recalled in one trial (10 words) and it ranges from 0 to 10. Pre-post trial changes in test results among the experimental group was compared with pre-post changes among the control group using linear regression models. (no drop out reported and therefore no need to use mixed effects models or MMRM)
Time Frame: 6 weeks (primary endpoint) from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of words
Arm/Group | Active Social Engagement Group | Control Group
Number analyzed (Participants) | 41 | 42
Number of words | -0.20 (1.72) | -0.19 (2.12)
Statistical Analysis 1: Comparison: Active Social Engagement Group vs Control Group; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.92, Regression, Linear; Mean Difference (Final Values) = -0.04, Standard Error of Mean 0.43 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Active Social Engagement Group vs Control Group; Analysis 2: CDR 0 (n=49); Test type: Equivalence — [test comment as in outcome 2, analysis 2]; p = 0.92, Regression, Linear; Mean Difference (Final Values) = 0.06, Standard Error of Mean 0.61 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Active Social Engagement Group vs Control Group; Analysis 3: CDR 0.5 (n=34); Test type: Equivalence — [test comment as in outcome 2, analysis 2]; p = 0.94, Regression, Linear; Mean Difference (Final Values) = -0.05, Standard Error of Mean 0.62 — [estimate comment as in outcome 1, analysis 1]

6. Primary Outcome: Changes in Trail Making Test A Scores (Post-study Test Score - Baseline Test Score)
Description: In Trail Making test A, the subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy within 150 seconds. Time to complete is used here. Pre-post trial changes in test results among the experimental group are compared with pre-post changes among the control group using linear regression models. (no drop out reported and therefore no need to use mixed effects models or MMRM). Larger changes mean subjects got slower to complete the test at the post-trial assessment. Negative changes indicates subjects completed the test faster at the post-trial assessment.
Time Frame: 6 weeks (primary endpoint) from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Active Social Engagement Group | Control Group
Number analyzed (Participants) | 41 | 42
Seconds | -2.80 (15.25) | -0.85 (9.51)
Statistical Analysis 1: Comparison: Active Social Engagement Group vs Control Group; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.46, Regression, Linear; Mean Difference (Final Values) = -2.11, Standard Error of Mean 2.84 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Active Social Engagement Group vs Control Group; Analysis 2: CDR 0 (n=49); Test type: Equivalence — [test comment as in outcome 2, analysis 2]; p = 0.61, Regression, Linear; Mean Difference (Final Values) = -1.07, Standard Error of Mean 2.08 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Active Social Engagement Group vs Control Group; Analysis 3: CDR 0.5 (n=34); Test type: Equivalence — [test comment as in outcome 2, analysis 2]; p = 0.80, Regression, Linear; Mean Difference (Final Values) = -1.66, Standard Error of Mean 6.42 — [estimate comment as in outcome 1, analysis 1]

7. Primary Outcome: Changes in Trail Making Test B Scores (Post-study Test Score - Baseline Test Score)
Description: In Trail Making test B, the subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy within 300 seconds. In Test B, the circles include both numbers (1 - 13) and letters (A - L). Time to complete is used here. Pre-post trial changes in test results among the experimental group are compared with pre-post changes among the control group using linear regression models. (no drop out reported and therefore no need to use mixed effects models or MMRM). Larger changes mean subjects got slower to complete the test at the post-trial assessment. Negative changes indicates subjects completed the test faster at the post-trial assessment.
Time Frame: 6 weeks (primary endpoint) from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Active Social Engagement Group | Control Group
Number analyzed (Participants) | 41 | 42
Seconds | -10.18 (29.32) | -14.65 (46.85)
Statistical Analysis 1: Comparison: Active Social Engagement Group vs Control Group; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.72, Regression, Linear; Mean Difference (Final Values) = 3.25, Standard Error of Mean 8.88 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Active Social Engagement Group vs Control Group; Analysis 2: CDR 0 (n=49); Test type: Equivalence — [test comment as in outcome 2, analysis 2]; p = 0.84, Regression, Linear; Mean Difference (Final Values) = 2.26, Standard Error of Mean 11.10 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Active Social Engagement Group vs Control Group; Analysis 3: CDR 0.5 (n=34); Test type: Equivalence — [test comment as in outcome 2, analysis 2]; p = 0.40, Regression, Linear; Mean Difference (Final Values) = 12.39, Standard Error of Mean 14.40 — [estimate comment as in outcome 1, analysis 1]

8. Primary Outcome: Changes in the Stroop Color and Word Test (Stroop Test C) Scores (Post-study Test Scores - Baseline Test Scores)
Description: In the Stroop test, subjects are required to read three different pages of stimuli in a designated time as quickly as possible. First, the individual is asked to name a series of colored squares (Color Naming task, Stroop Test A). Second, the individual is asked to read color words (Word Reading task, Stroop Test B). The final task is the Color-Word Naming task (Stroop Test C) on which the individual is shown the names of colors printed in conflicting ink colors (e.g., the word "red" in blue ink) and is asked to name the color of the ink rather than the word. Each test (A, B, C) is administered for 45 seconds. The number of words correctly named for the Stroop Test C was used here. The maximum score of this test is 100 (range: 0 - 100). The higher score indicates better functions. The changes (post-study - baseline test scores) among the experimental group are compared with those among the control group. The higher change scores mean improved function.
Time Frame: 6 weeks (primary endpoint) from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of words correctly named
Arm/Group | Active Social Engagement Group | Control Group
Number analyzed (Participants) | 41 | 42
Number of words correctly named | 0.34 (3.88) | 1.14 (4.29)
Statistical Analysis 1: Comparison: Active Social Engagement Group vs Control Group; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.38, Regression, Linear; Mean Difference (Final Values) = -0.81, Standard Error of Mean 0.91 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Active Social Engagement Group vs Control Group; Analysis 2: CDR 0 (n=49); Test type: Equivalence — [test comment as in outcome 2, analysis 2]; p = 0.39, Regression, Linear; Mean Difference (Final Values) = -1.12, Standard Error of Mean 1.31 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Active Social Engagement Group vs Control Group; Analysis 3: CDR 0.5 (n=34); Test type: Equivalence — [test comment as in outcome 2, analysis 2]; p = 0.59, Regression, Linear; Mean Difference (Final Values) = -0.68, Standard Error of Mean 1.26 — [estimate comment as in outcome 1, analysis 1]

9. Primary Outcome: Changes in Cogstate Computerized Test: Detection Test (Post-study Test Score - Baseline Test Score)
Description: In detection test, the on-screen instructions ask: "Has the card turned over?". A playing card is presented face down in the center of the screen. The card flips over so it is face up. As soon as the card flips over the participant must press "Yes". The participant is encouraged to work as quickly as they can and be as accurate as possible.Speed of performance (mean of the log10 transformed reaction times for correct responses) is used here. Pre-post trial changes in test results among the experimental group were compared with pre-post changes among the control group using linear regression models. (no drop out reported and therefore no need to use mixed effects models or MMRM). Larger changes mean subjects got slower in reaction at the post-trial assessment. Negative changes indicates subjects got faster in reaction at the post-trial assessment.
Time Frame: 6 weeks (primary endpoint) from baseline
Population: as for outcome 1
Measure: Mean (Standard Error); unit: log 10 milliseconds
Arm/Group | Active Social Engagement Group | Control Group
Number analyzed (Participants) | 41 | 42
log 10 milliseconds | 0.016 (0.091) | 0.065 (0.113)
Statistical Analysis 1: Comparison: Active Social Engagement Group vs Control Group; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.03, Regression, Linear; Mean Difference (Final Values) = -0.05, Standard Error of Mean 0.02 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Active Social Engagement Group vs Control Group; Analysis 2: CDR 0 (n=49); Test type: Equivalence — [test comment as in outcome 2, analysis 2]; p = 0.24, Regression, Linear; Mean Difference (Final Values) = -0.03, Standard Error of Mean 0.03 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Active Social Engagement Group vs Control Group; Analysis 3: CDR 0.5 (n=34); Test type: Equivalence — [test comment as in outcome 2, analysis 2]; p = 0.04, Regression, Linear; Mean Difference (Final Values) = -0.09, Standard Error of Mean 0.04 — [estimate comment as in outcome 1, analysis 1]

10. Primary Outcome: Changes in Cogstate One Back Accuracy (Post-study Test Score - Baseline Test Score)
Description: In this test, the on-screen instructions ask: "Is the previous card the same?". A playing card is presented face up in the center of the screen. The participant must decide whether the card is the same as the previous card. If the card is the same the participant should press "Yes", and if it is not the same the participant should press "No". The participant is encouraged to work as quickly as they can and be as accurate as possible. Accuracy of performance (arcsine transformation of the square root of the proportion of correct responses) is reported here. Pre-post trial changes in test results among the experimental group will be compared with pre-post changes among the control group using linear regression models. (no drop out reported and therefore no need to use mixed effects models or MMRM). Larger changes mean the score improved at the post trial assessment.
Time Frame: 6 weeks (primary endpoint) from baseline
Population: as for outcome 1
Measure: Mean (Standard Error); unit: arcsine transformed values (see above)
Arm/Group | Active Social Engagement Group | Control Group
Number analyzed (Participants) | 41 | 42
arcsine transformed values (see above) | 0.049 (0.246) | 0.062 (0.168)
Statistical Analysis 1: Comparison: Active Social Engagement Group vs Control Group; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.65, Regression, Linear; Mean Difference (Final Values) = -0.02, Standard Error of Mean 0.05 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Active Social Engagement Group vs Control Group; Analysis 2: CDR 0 (n=49); Test type: Equivalence — [test comment as in outcome 2, analysis 2]; p = 0.64, Regression, Linear; Mean Difference (Final Values) = 0.02, Standard Error of Mean 0.05 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Active Social Engagement Group vs Control Group; Analysis 3: CDR 0.5 (n=34); Test type: Equivalence — [test comment as in outcome 2, analysis 2]; p = 0.42, Regression, Linear; Mean Difference (Final Values) = -0.08, Standard Error of Mean 0.10 — [estimate comment as in outcome 1, analysis 1]

11. Primary Outcome: Changes in Cogstate Two Back Accuracy (Post-study Test Score - Baseline Test Score)
Description: In this test, the on-screen instructions ask: "Is the card the same as that shown two cards ago?". A playing card is presented face up in the center of the screen. The participant must decide whether the card is the same as the card shown two cards previously. If the card is the same the participant should press "Yes", and if it is not the same the participant should press "No". The participant is encouraged to work as quickly as they can and be as accurate as possible. Accuracy of performance (arcsine transformation of the square root of the proportion of correct responses) is reported here. Pre-post trial changes in test results among the experimental group will be compared with pre-post changes among the control group using linear regression models. (no drop out reported and therefore no need to use mixed effects models or MMRM)
Time Frame: 6 weeks (primary endpoint) from baseline
Population: as for outcome 1
Measure: Mean (Standard Error); unit: arcsine transformed values (see above)
Arm/Group | Active Social Engagement Group | Control Group
Number analyzed (Participants) | 41 | 42
arcsine transformed values (see above) | 0.020 (0.151) | 0.048 (0.209)
Statistical Analysis 1: Comparison: Active Social Engagement Group vs Control Group; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.45, Regression, Linear; Mean Difference (Final Values) = -0.03, Standard Error of Mean 0.45 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Active Social Engagement Group vs Control Group; Analysis 2: CDR 0 (n=49); Test type: Equivalence — [test comment as in outcome 2, analysis 2]; p = 0.93, Regression, Linear; Mean Difference (Final Values) = 0.004, Standard Error of Mean 0.05 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Active Social Engagement Group vs Control Group; Analysis 3: CDR 0.5 (n=34); Test type: Equivalence — [test comment as in outcome 2, analysis 2]; p = 0.40, Regression, Linear; Mean Difference (Final Values) = -0.07, Standard Error of Mean 0.08 — [estimate comment as in outcome 1, analysis 1]

12. Primary Outcome: Changes in CAMCI Total Score (Post-study Test Score - Baseline Test Score)
Description: Computer Assessment of Mild Cognitive Assessment (CAMCI) is a battery of computerized tasks to assess cognitive performance, developed by the Psychology Software Tools. The software provides standardized score (z-score) based on subject's age, sex and education.* The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean. Higher Z-score means better cognitive function. A positive change in Z-scores here indicates a favorable outcome. Total score (global cognitive function measure) is used here. Pre-post trial changes in test results among the experimental group are compared with pre-post changes among the control group using linear regression models. (no drop out reported and therefore no need to use mixed effects models or MMRM)
  *: Saxton J, Morrow L, Eschman A, Archer G, Luther J, Zuccolotto A. Computer assessment of mild cognitive impairment. Postgrad Med. 2009;121(2):177-85.
Time Frame: 6 weeks (primary endpoint) from baseline
Population: as for outcome 1
Measure: Mean (Standard Error); unit: z-score (standardized score)
Arm/Group | Active Social Engagement Group | Control Group
Number analyzed (Participants) | 41 | 42
z-score (standardized score) | 0.098 (0.394) | 0.182 (0.360)
Statistical Analysis 1: Comparison: Active Social Engagement Group vs Control Group; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.30, Regression, Linear; Mean Difference (Final Values) = -0.09, Standard Error of Mean 0.09 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Active Social Engagement Group vs Control Group; Analysis 2: CDR 0 (n=49); Test type: Equivalence — [test comment as in outcome 2, analysis 2]; p = 0.75, Regression, Linear; Mean Difference (Final Values) = 0.03, Standard Error of Mean 0.10 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Active Social Engagement Group vs Control Group; Analysis 3: CDR 0.5 (n=34); Test type: Equivalence — [test comment as in outcome 2, analysis 2]; p = 0.12, Regression, Linear; Mean Difference (Final Values) = -0.24, Standard Error of Mean 0.15 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Approximately eighteen weeks.
Description: Consistent with clinicaltrials.gov.
Arm/Group | Control Group | Active Soocial Engagement Group
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/41
Other Adverse Events (participants affected / at risk) | 0/42 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No